CLINICAL TRIAL: NCT05761145
Title: Relationship Between Sphingo-lipotoxicity and Trans-differentiation of Adipose Tissue: Cross-sectional Study in Subjects With Different Dysmetabolic Severity
Brief Title: Sphingo-lipotoxicity and Trans-differentiation of Adipose Tissue in Obesity (SFINGOTRANS)
Acronym: SFINGOTRANS
Status: Completed | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 01C126
Record Dates: First submitted 2023-02-27; First posted 2023-03-09 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Obesity; Healthy
Keywords: Obesity; Normals; Adipose tissue; Sphyngolipids; Metabolic syndrome
MeSH Terms: conditions — Obesity; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and serum samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cases - obese with metabolic syndrome: Obese subjects with metabolic syndrome
  Interventions: Diagnostic Test: Blood sample collection
- Cases - obese without metabolic syndrome: Obese subjects without metabolic syndrome
  Interventions: Diagnostic Test: Blood sample collection
- Controls: Normal weight subjects
  Interventions: Diagnostic Test: Blood sample collection

INTERVENTIONS:
Diagnostic Test: Blood sample collection — Blood sample collection

SUMMARY:
After recruiting a population of subjects with different metabolic severity (subjects of normal weight and obese patients with and without metabolic syndrome), the objectives of the present research will be:

1. determine leukocyte mRNA levels of Cidea (gene associated with BAT functional status), Hoxc9 (gene associated with browning of WAT) and Cpt1a (gene associated with β-oxidation of fatty acids in both tissues, i.e. BAT and WAT) (secondary endpoint);
2. to determine energy expenditure with indirect calorimetric technique, body temperature and circulating catecholamine levels, which will be correlated to leukocyte levels of Cidea, Hoxc9 and Cpt1a mRNA (secondary endpoint);
3. determine the plasma levels of an extensive panel of sphingolipids, including in particular ceramides and sphingosine-1-phosphate which, by exerting a lipotoxic, lipoinflammatory and anti-adipogenic effect, will be correlated to the leukocyte levels of Cidea, Hoxc9 mRNA and Cpt1a (primary endpoint);
4. determine the erythrocyte, leukocyte and platelet levels of sphingolipids which, acting as peripheral biomarkers of cardiometabolic dysfunction (e.g., atherogenesis, thromboembolism, arterial hypertension, insulin resistance, low-grade chronic inflammation, etc.), could phenotypically identify patients with increased cardiovascular risk (e.g., obese patients with or without metabolic syndrome) (secondary endpoint).

Hypothesis: the existence of a relationship between sphingohypotoxicity and transdifferentiation of adipose tissue and a combination of sphingolipids (plasma/erythrocyte/platelet/leukocyte) and gene regulators (WAT/BAT-related) which, with sensitivity and specificity, is associated with diagnosis of metabolic syndrome.

DETAILED DESCRIPTION:
Materials and methods Patients: 90 adults of both sexes will be recruited, of whom 30 of normal weight (age: 18-50 years; BMI < 25 kg/m2), 30 obese without metabolic syndrome (age: 18-35 years; BMI > 35 kg/m2) and 30 obese with metabolic syndrome (age: 18-35 years; BMI > 35 kg/m2), according to the 2009 IDF criteria. Subjects of normal weight will be recruited from medical/paramedical staff, while obese patients from hospitalized at the Division of Metabolic Diseases, Istituto Auxologico Italiano, Piancavallo (VB), Italy, for a 3-week multidisciplinary weight reduction program (BWRP), which includes low-calorie diet, physical exercise, psychological support and nutrition education.

Subjects with other pathologies other than obesity will be excluded from the study, including those treated with anticoagulant and antiplatelet drugs, since the evaluation of intraplatelet levels of sphingolipids will be foreseen.

In basal conditions, the main anthropometric data will be collected (weight, height, waist circumference, hip circumference, BMI), body composition will be evaluated with a bioimpedance technique, the main cardiovascular parameters will be recorded (blood pressure and heart rate), a calorimetric examination will be performed, collection of body temperature (morning and evening), request of the environmental temperature to which one is generally exposed during the day and determined, with automated clinical biochemistry techniques, the following biochemical parameters: glucose, total cholesterol, triglycerides, LDL, HDL, fatty acids non-esterified, insulin, glycated Hb, catecholamines and C-reactive protein.

Determination of the lipidomic profile in plasma and cell extracts A lipidomics will be performed in plasma and in cellular extracts from erythrocytes, leukocytes and platelets. The levels of the individual analytes will be determined with a technologically advanced analytical instrumentation, consisting of a triple quadruple hybrid mass spectrometer with linear ion trap (QTRAP 5500, AB Sciex), interfaced with an ultra-high performance liquid chromatograph (UHPLC).

Plasma and cellular levels of the following sphingolipids will be measured: ceramides and dihydroceramides from C16 to C24, including 2 unsaturated ones (C18:1 and C24:1), the sphingomyelins (those from C16 to C24 and the one C24:1), sphingosine, sphinganine , sphingosine-1-phosphate and sphinganine-1-phosphate.

Determination of leukocyte mRNA levels of gene regulators From an aliquot containing leukocytes, stored ad hoc, the total mRNA will be extracted and, with RT/PCR technique, the leukocyte mRNA levels of the following genes will be determined: Cidea, Hoxc9 and Cpt1a.

ELIGIBILITY:
Inclusion Criteria (obese subjects):

- obesity (BMI > 35 kg/m2)

Inclusion criteria (healthy controls):

- BMI < 25 kg/m2

Exclusion Criteria:

- patients/controls treated with anticoagulant and antiplatelet drugs

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Obese patients (BMI > 35 kg/m2) and age- and sex-matched healthy controls (normal weighted)
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2022-03-23 (Actual); Study Completion 2022-03-23 (Actual)

PRIMARY OUTCOMES:
Evaluation of sphingolipids | Baseline
  Determination of an extensive panel of sphingolipids, including ceramides and sphingosine-1-phosphate which, by exerting a lipotoxic, lipoinflammatory and anti-adipogenic effect, are correlated to the leukocyte levels of Cidea, Hoxc9 mRNA and Cpt1a

SECONDARY OUTCOMES:
Determination of leukocyte mRNA levels of Cidea and Cpt1a | Baseline
  determination of leukocyte mRNA levels of Cidea (gene associated with BAT functional status), Hoxc9 (gene associated with browning of WAT) and Cpt1a (gene associated with β-oxidation of fatty acids in both tissues, i.e. BAT and WAT)
Determination of the erythrocyte, leukocyte and platelet levels of sphingolipids | Baseline
  Determination of the erythrocyte, leukocyte and platelet levels of sphingolipids which, acting as peripheral biomarkers of cardiometabolic dysfunction (e.g., atherogenesis, thromboembolism, arterial hypertension, insulin resistance, low-grade chronic inflammation, etc.), could phenotypically identify patients with increased cardiovascular risk (e.g., obese patients with or without metabolic syndrome)

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano, Site Piancavallo, Oggebbio, Verbania, Italy